CLINICAL TRIAL: NCT00257790
Title: Tobramycin én Gang Daglig Mot Tre Ganger Daglig, Gitt Med Benzylpenicillin, Til Pasienter Med nøytropen Feber
Brief Title: The Tobramycin Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The National Institute of Health, Oslo (Unknown); Ullevaal University Hospital (Other); Sorlandet Hospital HF (Other Government); Sykehuset Buskerud (Unknown); Sentralsjukehuset i Rogaland (Unknown); Sykehuset Innlandet HF (Other); Sentralsjukehuset i Hedemark (Unknown); The Hospital of Vestfold (Other); Sykehuset Asker og Baerum (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tobrax1; 01-06850; 8560; 2016
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-11

CONDITIONS: Neutropenia; Fever; Cancer
Keywords: Fever; Neutropenia; Tobramycin; Aminoglycoside; Penicillin
MeSH Terms: conditions — Neutropenia; Fever; Neoplasms

INTERVENTIONS:
Drug: Tobramycin once a day

SUMMARY:
Evaluate if tobramycin given once a day is at least as efficacious as the traditional tobramycin given three times a day, given with penicillin G, til patients with febrile neutropenia.

DETAILED DESCRIPTION:
Prospective randomized Norwegian multicenter clinical trial (11 hospitals) comparing tobramycin given once a day (new regimen) vs. three times a day (current regimen), with penicillin G, to cancer patients with febrile neutropenia. Tobramycin half life and postantibiotic effect is at best 12 hours. It has been questioned if tobramycin once a day is safe in patients with low levels of granulocytes when it is given with a drug like penicillin G which is not covering Gram-negative rods. Treatment of febrile neutropenia with penicillin G and an aminoglycoside is standard of care in Norway, and it is probably a regimen that is promoting antimicrobial resistance less than a broad spectrum beta-lactam.

Cancer patients 16-70 with febrile neutropenia and signed informed consent could be randomized. Exclusion criteria were allergy to study medications, increased creatinine/renal failure, massive ascites, multiple myeloma, treatment with cis-platinum, recent therapy with aminoglycoside (4 weeks) or other antibiotics (4 days), hemodynamically unstable patients, pregnant and nursing patients.

Patients were stratified into three groups: Leukemia patients receiving intensive chemotherapy, lymphoma patients receiving high dose chemotherapy with autologous stem-cell support and other cancer patients.

Patients were randomized to either tobramycin once or three times a day. Once the patient was randomized and the first antibiotic dose was given, further antibiotic therapy was up to the patient's doctor's discretion (not blinded). Everybody received tobramycin 6 mg/kg/day and penicillin 5 mill. IE four times a day.

The patients were followed until all antibiotic therapy was terminated. Clinical condition and laboratory test results at time of randomization (new fever) was registered. Response to therapy, reason for modification of therapy, mortality, duration of neutropenia, maximum creatinine level, tobramycin serum concentrations, microbiological findings and total antibiotic consumption were registered.

After external monitoring of all the data the results are currently being made up and will be available for publication in 2006.

This trial has been conducted independently of the pharmaceutical industry. Grants have been received from The Norwegian Radium Hospital research fund, The Regional Health Authorities and The Norwegian Society for Infectious Diseases.

ELIGIBILITY:
Febrile neutropenia Cancer Adult (16-70) Signed informed consent

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2001-09; Study Completion 2005-03

PRIMARY OUTCOMES:
Resolution of fever and signs of infection without modification of the antibiotic regimen

SECONDARY OUTCOMES:
Hours to defervescence
Days to treatment failure
30 days mortality
Nephrotoxicity
Other side effects
Pharmacokinetics of tobramycin in febrile neutropenic patients
Total antibiotic consumption
Cost-benefit of giving tobramycin once a day vs three times a day

CONTACTS AND LOCATIONS:
Overall Officials: Dag Torfoss, MD, Principal Investigator — Oslo University Hospital